CLINICAL TRIAL: NCT05648058
Title: Role of Nefopam in Rituximab Transfusion Reaction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry Of Health / Nineveh Health Directorate (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: nefopam with rituximab
Record Dates: First submitted 2022-12-04; First posted 2022-12-13 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Nefopam
MeSH Terms: interventions — Nefopam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nefopam (Experimental): administration of intravenous nefopam to prevent Rituximab Transfusion Reaction
  Interventions: Drug: Nefopam ampule
- diphenhydramine (Active Comparator): administration of intravenous diphenhydramine to prevent Rituximab Transfusion Reaction
  Interventions: Drug: diphenhydramine ampule

INTERVENTIONS:
Drug: Nefopam ampule — nefopam ampule 50 mg
  Other Names: ACUPAN
  Arms: nefopam
Drug: diphenhydramine ampule — diphenhydramine ampule 10 mg
  Other Names: Allermine
  Arms: diphenhydramine

SUMMARY:
the patients will be taken nefopam ampule 50 mg before rituximab in the first group while the second group will be taken diphenhydramine ampule 10 mg before rituximab in the second group

DETAILED DESCRIPTION:
the two groups will be taken standard therapy (hydrocortisone vial 100 mg and acetaminophen 1000 mg) 30 min before rituximab

ELIGIBILITY:
Inclusion Criteria:

* 18 - 80 years old male and female will be taken rituximab

Exclusion Criteria:

* less than 18 years old more than 80 years old diabetic patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2023-10-20 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
transfusion reaction | 30 min
  fever, riger, rash, chills, pruritus and bronchospasm

CONTACTS AND LOCATIONS:
Overall Officials: moataz alani, Study Chair — Ministry Of Health / Nineveh Health Directorate

IPD SHARING:
Plan to Share IPD: No